CLINICAL TRIAL: NCT00197756
Title: Vitamins, Breastmilk HIV Shedding, and Child Health
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Eduardo Villamor, MD, DrPH, Harvard School of Public Health
Other Study IDs: HD45134
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2009-08-21 (Estimated); Status verified 2009-08

CONDITIONS: Maternal and Child Health Outcomes
Keywords: HIV; Breastfeeding; Vitamins; Tanzania; Children
MeSH Terms: conditions — Breast Feeding | interventions — Vitamin A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breast milk samples collected from breast at delivery and at 3 month intervals thereafter.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Vitamin A: Participants in the in the parent study who had been randomized to receive either Vitamin A alone or multivitamins including vitamin A.
  Interventions: Dietary Supplement: Vitamin A alone
- No Vitamin A: Participants in the parent study who were randomized to receive either multivitamins excluding vitamin A, or placebo.
  Interventions: Dietary Supplement: Multivitamins excluding vitamin A; Dietary Supplement: multivitamins including vitamin A; Other: Placebo
- Multivitamins: Participants in the parent study who were randomized to receive multivitamins including vitamin A or multivitamins excluding vitamin A
  Interventions: Dietary Supplement: Vitamin A alone; Dietary Supplement: Multivitamins excluding vitamin A; Dietary Supplement: multivitamins including vitamin A
- No Multivitamins: Participants from the parent study who had been randomized to vitamin A alone or placebo
  Interventions: Dietary Supplement: Vitamin A alone; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin A alone — 30 mg beta-carotene plus 5000 IU preformed vitamin A) taken orally once per during pregnancy and lactation
  Groups: Multivitamins; No Multivitamins; Vitamin A
Dietary Supplement: Multivitamins excluding vitamin A — 30 mg thiamine, 20 mg riboflavin, 20 mg B-6, 100 mg niacin, 50 ug vitamin B-12, 500 mg vitamin C, 30 mg vitamin E, 0.8 mg folic acid taken orally once per day during pregnancy and lactation
  Groups: Multivitamins; No Vitamin A
Dietary Supplement: multivitamins including vitamin A — 20 mg thiamine, 20 mg riboflavin, 25 mg vitamin B6, 100 mg niacin, 50 ug vitamin B12, 500 mg vitamin C, 30 mg vitamin E, and 0.8 mg folic acid taken once per day orally during pregnancy and lactation
  Groups: Multivitamins; No Vitamin A
Other: Placebo — Placebo pill taken orally once per day during pregnancy and lactation
  Groups: No Multivitamins; No Vitamin A

SUMMARY:
The purpose of this study is to analyze stored samples and data collected during the conduct of the study "A Trial of Vitamins in HIV Progression and Transmission" (HD32257). The aims are to examine the effect of vitamin supplementation on HIV infected women during pregnancy on a number of parameters in breastmilk.

DETAILED DESCRIPTION:
The purpose of this study is to analyze stored samples and data collected during the conduct of the study "A Trial of Vitamins in HIV Progression and Transmission" (HD32257). The aims are to examine the effect of vitamin supplementation on HIV infected women during pregnancy

ELIGIBILITY:
This study is analyzing samples previously collected from the study "A Trial of Vitamins in HIV Progression and Transmission" (HD32257).

The inclusion criteria in this study was:

* HIV infected women presenting to antenatal care between 12 and 27 weeks of gestation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data and samples used in this study are from HIV-infected pregnant women who participated in the "Trial of Vitamins in HIV Transmission and Progression". Between 1995 and 1997, 1,078 African, HIV positive women who were between gestatopm weeks 12 and 27 were recruited. They were followed until August 2003. This study was conducte among 771 of these women, for whom breast milk samples were available at delivery. There were no differences in baseline characteristics between this subset and the originally randomized group of 1,069.
Sampling Method: Non-Probability Sample
Enrollment: 771 (Actual)
Dates: Start 2004-09; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
cell-free viral load and/or cell-associated proviral load in breast milk | Delivery, 3 months, and 6 months after delivery
concentration of vitamins A, B12, and E in breast milk | Delivery, 3 months, and 6 months post-delivery
subclinical mastitis | Delivery, 3 months, and 6 months after delivery

SECONDARY OUTCOMES:
post-natal mother-to-child transmission of HIV | Delivery, 3 months, and 6 months post-delivery
infant mortality and morbidity from diarrhea | Delivery, 3 months and 6 months after delivery
a.) CCR5 expression in differentiating monocytes and differentiated monocyte-derived macrophages | N/A (in vitro experiment)
HIV-1 replication in differentiating monocytes acutely infected with a subtype C HIV-1 clone, differentiated non-dividing MDMs acutely infected with the HIV-1 MJ4 clone, and differentiated non-dividing MDMs chronically infected with the HIV-1 MJ4 clone. | N/A (in vitro experiment)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Villamor, MD,DrPH, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (1):
- Harvard School of Public Health, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Villamor E, Koulinska IN, Aboud S, Murrin C, Bosch RJ, Manji KP, Fawzi WW. Effect of vitamin supplements on HIV shedding in breast milk. Am J Clin Nutr. 2010 Oct;92(4):881-6. doi: 10.3945/ajcn.2010.29339. Epub 2010 Aug 25. PMID 20739426
- [Derived] Webb AL, Aboud S, Furtado J, Murrin C, Campos H, Fawzi WW, Villamor E. Effect of vitamin supplementation on breast milk concentrations of retinol, carotenoids and tocopherols in HIV-infected Tanzanian women. Eur J Clin Nutr. 2009 Mar;63(3):332-9. doi: 10.1038/sj.ejcn.1602929. Epub 2007 Oct 17. PMID 17940544